CLINICAL TRIAL: NCT04347122
Title: Tranexamic Acid in Radical Resection and Endoprosthetic Reconstruction: A Randomized Controlled Trial
Brief Title: Tranexamic Acid in Radical Resection and Endoprosthetic Reconstruction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment stalled
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Kyle Sweeney, MD, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00144738
Record Dates: First submitted 2020-04-06; First posted 2020-04-15 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Musculoskeletal Cancer; Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of four groups. One group is the bony tumor treated with TXA, second group is the bony tumor treated without TXA, third group is the soft tissue sarcoma treated with TXA, and the fourth group is soft tissue sarcoma treated without TXA.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Bony tumor treated with Tranexamic acid (TXA) (Active Comparator): This group of participants will undergo a bony tumor resection of the femur or proximal tibia and endoprosthetic reconstruction with TXA.
  Interventions: Drug: Tranexamic Acid (TXA)
- Bony tumor treated without TXA (No Intervention): This group of participants will undergo a bony tumor resection of the femur of proximal tibia and endoprosthetic reconstruction.
- Soft tissue sarcoma treated with Tranexamic Acid (TXA) (Active Comparator): This group of participants will undergo soft tissue sarcoma resection of the lower extremity with TXA
  Interventions: Drug: Tranexamic Acid (TXA)
- Soft tissue sarcoma treated without TXA (No Intervention): This group of participants will undergo soft tissue sarcoma resection of the lower extremity.

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — Intervention groups will receive TXA 1g TXA IVPB 10 minutes prior to incision and a second dose of 1g IVPB at the time of closure.
  Arms: Bony tumor treated with Tranexamic acid (TXA); Soft tissue sarcoma treated with Tranexamic Acid (TXA)

SUMMARY:
This study intends to determine if any correlation exists between administration of TXA or not to musculoskeletal oncology patients undergoing endoprosthetic reconstruction and blood loss and blood transfusion rates.

DETAILED DESCRIPTION:
Resection of bony and soft tissue tumors with endoprosthetic reconstruction often presents a significant risk of perioperative blood loss requiring transfusion. Tranexamic acid (TXA) is an antifibrinolytic that is commonly used to reduce blood loss in orthopedic procedures, most often arthroplasty. The aim of this study is to determine in a randomized controlled fashion if there is any difference in perioperative blood loss and blood transfusion rates when TXA is used compared to when it is not used in patients undergoing radical resection of bone and soft tissue sarcomas with endoprosthetic reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing wide resection of a malignant bony tumor of the lower extremity with endoprosthetic reconstruction.
* Patients undergoing a resection of soft tissue sarcoma measuring > 5cm.

Exclusion Criteria:

* Patients undergoing revision endoprosthetic reconstruction
* Patients with known coagulopathy
* Known history of DVT or embolic disease
* Benign tumors
* Patients with allergy to TXA
* Those refusing blood products
* Those concurrently on anti-coagulant therapy
* Pregnant and/or nursing women
* Vulnerable populations as defined by the KUMC IRB

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Sweeney, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bony Tumor w/ TXA Group: bony tumor that will receive TXA
- Bony Tumor no TXA Group: bony tumor with no TXA treatment
- Soft Tissue Tumor w/ TXA Group: soft tissue tumor that will receive TXA
- Soft Tissue Tumor With no TXA Group: soft tissue tumor with no TXA
Period: Overall Study
Arm/Group | Bony Tumor w/ TXA Group | Bony Tumor no TXA Group | Soft Tissue Tumor w/ TXA Group | Soft Tissue Tumor With no TXA Group
Started | 0 | 3 | 3 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 3 | 6
Not completed — Physician Decision | 0 | 3 | 3 | 6

BASELINE CHARACTERISTICS:
Population: Enrollment was terminated, study was closed due to low enrollment, therefore no data were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bony Tumor Treated With Tranexamic Acid (TXA) | Bony Tumor Treated Without TXA | Soft Tissue Sarcoma Treated With Tranexamic Acid (TXA) | Soft Tissue Sarcoma Treated Without TXA | Total
Number analyzed (Participants) | 0 | 3 | 3 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3 | 6 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 3 | 5
  Male | 0 | 2 | 2 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Blood Loss
Description: How much blood was lost during surgical process
Time Frame: During surgical procedure, 4 to 6 hours
Population: Bony tumor w/ TXA group had no participants
Measure: Mean (Full Range); unit: mL
Arm/Group | Bony Tumor w/ TXA Group | Bony Tumor no TXA Group | Soft Tissue Tumor w/ TXA Group | Soft Tissue Tumor With no TXA Group
Number analyzed (Participants) | 0 | 3 | 3 | 6
mL |  | 283 [250 to 350] | 700 [100 to 1800] | 416 [100 to 700]

ADVERSE EVENTS:
Time Frame: up to 3 days
Description: There were no subjects in Bony tumor w/ TXA group.
Groups:
- Bony Tumor w/ TXA Group; Soft Tissue Tumor w/ TXA Group: Participants received TXA
- Bony Tumor no TXA Group; Soft Tissue Tumor With no TXA Group: Participants did not receive TXA
Arm/Group | Bony Tumor w/ TXA Group | Bony Tumor no TXA Group | Soft Tissue Tumor w/ TXA Group | Soft Tissue Tumor With no TXA Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/3 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/0 | 0/3 | 0/3 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT04347122/Prot_SAP_003.pdf
  • Informed Consent Form (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT04347122/ICF_001.pdf